CLINICAL TRIAL: NCT00379353
Title: The Effects of Thalidomide on Symptom Clusters
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2005-0980
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Results first posted 2013-01-01 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; Anorexia; Fatigue; Thalidomide; Placebo
MeSH Terms: conditions — Anorexia; Fatigue | interventions — Thalidomide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: Thalidomide (Active Comparator): 100 mg capsules orally, once a day for 14 days
  Interventions: Drug: Thalidomide
- Group 2: Placebo (Placebo Comparator): Two placebo capsules orally, once a day for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Thalidomide — 100 mg capsules orally, once a day for 14 days.
  Arms: Group 1: Thalidomide
Drug: Placebo — Two placebo capsules orally, once a day for 14 days.
  Arms: Group 2: Placebo

SUMMARY:
The goal of this clinical research study is to learn if thalidomide can improve symptoms such as pain, fatigue,anxiety, poor appetite, depression, and sleep problems in patients with advanced cancer.

DETAILED DESCRIPTION:
Thalidomide is designed to change the immune system. It may also interfere with the development of tiny blood vessels that help support tumor growth.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will be asked about your cancer diagnosis, the drugs you are taking, and the symptoms you are having (for example, pain, fatigue, anxiety, depression, poor appetite, and sleep problems). Blood (about 2 tablespoons) will be drawn to measure protein levels in your blood.

Women who are able to have children must have a negative blood (about 1 tablespoon) pregnancy test 24 hours before beginning to receive thalidomide.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in toss of a coin) to one of 2 groups. You will have an equal chance of being placed in either of the 2 groups. You, the medical staff, and researchers will not know which group you have been assigned to.

Participants in Group 1, who are not on chemotherapy, will take 2 thalidomide capsules, by mouth, once a day for 14 days. Participants in Group 1, who are on chemotherapy, will take 1 thalidomide capsule, by mouth, once a day for 7 days, and then 2 thalidomide capsules, by mouth, once a day for 7 days.

Participants in Group 2, who are not on chemotherapy, will take 2 placebo capsules, by mouth, once a day for 7 days. Participants in Group 2, who are on chemotherapy, will take 1 placebo capsule, by mouth, once a day for 7 days, and then 2 placebo capsules, by mouth, once a day for 7 days. A placebo is a substance that looks like the study drug but has no active ingredients.

You will complete 7 questionnaires, which will take about 30-60 minutes to complete. You will also have blood drawn (about 2 tablespoons) to measure protein levels in your blood. You will also have your body weight measured and be asked about your normal food intake. Your body composition will be measured using measurements that include body weight and height, skin fold thickness using Lange calipers, and bioelectrical impedance using the Tanita body composition monitoring scale. This is a non-invasive method to measure total body water, total body fat, and total body lean mass. The Tanita scale is similar to a typical weight scale, although unlike a weight scale, the Tanita scale measures body composition. Researchers will measure how much energy your body uses while at rest.

Every week, women who are able to have children must have a negative blood (about 1 tablespoon) pregnancy test.

On Day 8 [± 3 days], you will complete 3 questionnaires. The 3 questionnaires include evaluation of your symptoms, fatigue level, and overall sense of well-being and should take about 30 minutes to complete.

On Day 15 [± 3 days] you will have a study visit. You will be asked questions about any side effects you may have experienced. You will be asked about any symptoms of pain, fatigue, nausea, depression, poor appetite, and/or sleep problems. You will be asked to complete 7 questionnaires which will take about 30-60 minutes to complete. You will also have your body weight measured and be asked about your normal food intake. Your body composition will be measured and researchers will measure how much energy your body uses while at rest. Blood (about 2 tablespoons) will be drawn to measure protein levels in your blood. All patients will be given the option to receive thalidomide until Day 30 [± 3 days].

If you decide not to take thalidomide on Days 15-30, you will be considered off-study. If you decide to take thalidomide on Days 15-30, you will remain on study until Day 30. On Day 30 [± 3 days], you will have end-of-study tests.

On Day 30 [± 3 days], you will have an end-of-study visit. You will be asked questions about any side effects you may have experienced. You will be asked about any symptoms of pain, fatigue, anxiety, depression, poor appetite, and/or sleep problems.

Blood (about 2 tablespoons) will be drawn to measure protein levels in your blood. You will be asked to complete 7 questionnaires which will take about 30-60 minutes to complete. You will also have your body weight measured and be asked about your normal food intake. Your body composition will be measured and researchers will measure how much energy your body uses while at rest.

If you develop intolerable side effects, you will be taken off study. Otherwise, you will be considered off-study on either Day 15 [± 3 days] or Day 30 [± 3 days]. Blood (about 1 tablespoon) will be drawn 2 weeks after thalidomide has been stopped to check for additional side effects.

You and your doctor will have the option to continue your taking thalidomide off-study. You will participate in the S.T.E.P.S.® (System for Thalidomide Education and Prescribing Safety) program. This will include an additional consent, education about preventing pregnancy while taking thalidomide, and completing surveys about following the rules of this program.

This is an investigational study. Thalidomide is FDA-approved and commercially available. Its use in this study, for this purpose, is investigational. Up to 62 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Have weight loss of > 5% within the last 6 months
2. Present with anorexia, fatigue and one of the following: anxiety, depression or sleep disturbances, during the preceding 24 hours, with an average intensity of each symptom >/= 3 on a scale of 0 to 10, in which 0=no symptom, and 10= the worst possible symptom.
3. Describe the symptoms as being present every day for a minimum of 2 weeks.
4. Have no clinical evidence of cognitive failure
5. Must be 18 years or older.
6. Expect to live at least >/= 4 weeks
7. Must have negative serum pregnancy test within 24 hours of study enrollment in women of childbearing potential. FDA criteria for the status of not of childbearing potential, hysterectomy, or menopausal for 24 consecutive months.
8. Understand and sign written informed consent.
9. Have no concurrent steroids with the exception of steroids used concurrently with chemotherapy as part of a regimen or to reduce nausea.
10. Willing and able to comply with S.T.E.P.S.[System for Thalidomide Education and Prescribing Safety]
11. Patient's Absolute neutrophil count (ANC) at time of study enrollment is >/= 750 mm (to be drawn within 14 days prior to registration)
12. May be on chemotherapy if at a stable dose. Targeted therapies or hormone therapies are permitted once patient has completed two weeks of treatment.

Exclusion Criteria:

1. Have major contraindication to thalidomide, i.e. hypersensitivity.
2. Present with National Cancer Institute (NCI) Common Toxicity Criteria Grade 3 or more peripheral neuropathy.
3. Are not able to complete the baseline assessment forms.
4. Are pregnant or lactating.
5. Patients with clinical history of seizures
6. Patients with an ANC of </= 750 at time of study enrollment will be excluded (to be drawn within 14 days prior to registration).
7. Patients with a history of Acquired Immune Deficiency Syndrome (AIDS), systemic lupus erythematous, or renal failure as defined by a serum creatinine of > 2.0 mg/dl at baseline will be excluded (to be drawn within 29 days prior to registration).
8. Patients on Revlimid (lenalidomide).
9. Patients on investigational chemotherapy/agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bruera, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 10/18/2006 through 10/27/2008. All participants recruited from UTMD Anderson Cancer Center.
Pre-assignment Details: The trial is now closed to new participant entry due to low accrual. Of the 31 participants recruited, 4 were not eligible for evaluation.
Period: Overall Study
Arm/Group | Group 1: Thalidomide | Group 2: Placebo
Started | 16 | 15
Completed | 5 | 9
Not Completed | 11 | 6
Not completed — Hospitalization | 3 | 3
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Death | 1 | 0
Not completed — Cardiac Tamponade | 1 | 0
Not completed — Non-compliance | 1 | 0
Not completed — Conflicting drug treatment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Thalidomide | Group 2: Placebo | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 4 | 4 | 8
Age Continuous [Median (Full Range); unit: years] | 60 [24 to 81] | 65 [49 to 81] | 60 [24 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31

OUTCOME MEASURES:

1. Secondary Outcome: Functional Assessment of Anorexia/Cachexia Therapy (FAACT)
Description: 12-item symptom-specific subscale of the FACT-G designed to measure participants' additional concerns about their anorexia/cachexia during the previous 7 days. Participant rates concerns from 0 to 4 (0= not at all, 4= very much), combined are the 12 items subscales for a total of 0 to 48 where the higher number would represent greater concern.
Time Frame: Baseline to Day 29
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Group 1: Thalidomide | Group 2: Placebo
Number analyzed (Participants) | 16 | 15
units on a scale
  Baseline | 22.5 [9 to 36] | 22.5 [19 to 32]
  Day 15 | 32 [13 to 38] | 28 [21 to 32]
  Day 29 | 25 [19 to 38] | 27 [22 to 39]

2. Secondary Outcome: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F)
Description: The FACIT-F consists of 27 general quality of life questions divided into 4 domains (physical, social, emotional and functional), plus a 13-item fatigue subscore. The participant rates the intensity of fatigue and its related symptoms on a scale of 0-4 (0= not at all, 4= very much) where the 13-item fatigue subscore totals are combined for a total of 0 to 52, with the higher number representing greater fatigue.
Time Frame: Baseline to Day 29
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Group 1: Thalidomide | Group 2: Placebo
Number analyzed (Participants) | 16 | 15
units on a scale
  Baseline | 21 [7 to 35] | 20 [15.5 to 25]
  Day 15 | 24.5 [4 to 39] | 24 [17 to 31]
  Day 29 | 16 [9 to 34] | 24 [18 to 32]

3. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) HADS-A (Anxiety)
Description: The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). The higher the score The higher the score, the more likely the patient is showing signs of anxiety and as a result may benefit from a counseling/supportive session.
Time Frame: Baseline to Day 29
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Group 1: Thalidomide | Group 2: Placebo
Number analyzed (Participants) | 16 | 15
units on a scale
  Baseline | 9 [2 to 16] | 7 [4 to 9]
  Day 15 | 9 [1 to 9] | 4 [2 to 10]
  Day 29 | 6 [5 to 10] | 6.5 [4.2 to 10]

4. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) HADS-D (Depression)
Description: The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). The higher the score, the more likely the patient is showing signs of depression and as a result may benefit from a counseling/supportive session.
Time Frame: Baseline to Day 29
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Group 1: Thalidomide | Group 2: Placebo
Number analyzed (Participants) | 16 | 15
units on a scale
  Baseline | 10 [4 to 17] | 8 [3 to 10]
  Day 15 | 8 [3 to 13] | 8.5 [3 to 12]
  Day 29 | 8 [4 to 17] | 6.59 [4.2 to 10]

5. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: PSQI measures the quality and patterns of sleep. It differentiates poor from good sleep by measuring subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. A participant indicates how frequently each item was experienced on a scale from 0 to 3. The 7 component scores are then summed to obtain a global sleep score that can range from 0 to 21. A score of >/= 5 indicates poor sleepers.
Time Frame: Baseline to Day 29
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Group 1: Thalidomide | Group 2: Placebo
Number analyzed (Participants) | 16 | 15
units on a scale
  Baseline | 9.5 [7.5 to 14.7] | 11 [5.2 to 15]
  Day 15 | 10.5 [5.25 to 12.7] | 8.5 [3.25 to 13.5]
  Day 29 | 8 [3 to 10] | 8 [4 to 12]

6. Primary Outcome: Change in Symptoms as Measured by Edmonton Symptom Assessment Scale (ESAS)
Description: ESAS assessment of appetite (symptom) where the severity at the time of assessment is rated from 0 to 10 on a numerical scale; with 0 meaning that the symptom is absent and 10 that it is the worst possible severity. Evaluated at baseline [± 3 days], 2 weeks[± 3 days] and 4 weeks [± 3 days]
Time Frame: Baseline to Day 29
Measure: Median (Full Range); unit: units on a scale
Groups:
- Thalidomide (Baseline); Thalidomide (Day 15); Thalidomide (Day 29): Thalidomide 100 mg capsules orally, once a day for 14 days.
- Placebo (Baseline); Placebo (Day 15); Placebo (Day 29): Two placebo capsules orally, once a day for 14 days.
Arm/Group | Thalidomide (Baseline) | Thalidomide (Day 15) | Thalidomide (Day 29) | Placebo (Baseline) | Placebo (Day 15) | Placebo (Day 29)
Number analyzed (Participants) | 16 | 16 | 16 | 15 | 15 | 15
units on a scale
  Pain | 3 [0 to 8] | 3 [0 to 10] | 4 [0 to 8] | 3 [2 to 5] | 6.5 [0 to 6.5] | 2.5 [2.5 to 3]
  Fatigue | 7 [2 to 8] | 5.5 [1 to 9] | 5 [2 to 6] | 6.5 [4.25 to 8] | 5 [2.5 to 5.5] | 5 [3.25 to 8]
  Appetite | 6 [3 to 10] | 4.5 [1 to 8] | 7 [0 to 10] | 6.5 [0 to 6.5] | 3 [2 to 7] | 5.5 [2.25 to 8]
  Depression | 6 [0 to 10] | 1.5 [0 to 7] | 2 [0 to 5] | 2.5 [0 to 4.7] | 2 [0 to 3] | 2 [0 to 3.75]

7. Secondary Outcome: Change in Body Composition as Measured by Body Mass Index (BMI)
Description: BMI, commonly used to measure overweight and obesity, is a measure of body fat based on a person's weight and height.
Time Frame: Baseline to Day 29
Measure: Median (Full Range); unit: kg/m^2
Arm/Group | Thalidomide (Baseline) | Thalidomide (Day 15) | Thalidomide (Day 29) | Placebo (Baseline) | Placebo (Day 15) | Placebo (Day 29)
Number analyzed (Participants) | 16 | 16 | 16 | 15 | 15 | 15
kg/m^2 | 21.1 [20.2 to 25.4] | 21.2 [20.75 to 23.8] | 23.4 [19.6 to 28.2] | 22.3 [19.4 to 26.9] | 23.7 [19.4 to 26.9] | 22.1 [19.1 to 26.9]

8. Secondary Outcome: Change in Serum Cytokines and Receptors
Description: Cytokines Levels of IL-1β and its receptor IL RA, IL-6 its receptor IL-6R, and TNF-α and its receptors (i.e. tumor necrosis factor receptor (TNFR)) of TNFR1, TNFR2, IL-10, IL-8(serum) measured at baseline, Days 15 and 29. Multiplex bead Immunoassay used to measure serum/plasma levels of IL-1, IL-6, TNF-α, IL-10, IL-8 and their receptors where assay sensitivity for the cytokines was 3-6 pg/mL. Serum IL-10, IL-1β, IL-1RA, IL-6R, sTNF-RI, sTNF-R2 were also analyzed using an enzyme-linked immunosorbent assay device. Lowering cytokine levels can decrease fatigue, increase appetite and decrease anxiety and depression.
Time Frame: Baseline to Day 15
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Thalidomide (Baseline) | Thalidomide (Day 15) | Placebo (Baseline) | Placebo (Day 15)
Number analyzed (Participants) | 16 | 16 | 15 | 15
pg/mL
  IL-6 | 54.1 [16.8 to 280.3] | 85 [18 to 140] | 76.4 [19.1 to 133] | -6.51 [-37.9 to 26.4]
  IL-1b | 0.52 [0.32 to 0.74] | 0.67 [0.29 to 2.77] | 0.83 [0.22 to 1.4] | 0.57 [0.43 to 0.68]
  IL1RA | 677 [501 to 784] | 290.7 [-901 to 515] | 579 [266 to 755] | 102.3 [-639.6 to 356.3]
  Tumor necrosis factor -a (TNF-a) | 18.2 [13.8 to 123.1] | 6.4 [-24.8 to 108.8] | 21.2 [17.8 to 37.1] | 6.24 [-12.8 to 14.6]
  IL-17 | 3.2 [1.75 to 39.7] | 9.2 [3.1 to 17] | 12.07 [4.3 to 122.6] | 11 [3.4 to 316.3]
  IL-8 | 36.1 [29.7 to 68.1] | 2.12 [-7.5 to 11.2] | 139.9 [54.1 to 289.1] | -3.7 [-20.9 to 50.3]
  IL-6R | 6264 [4321 to 30159] | 5446 [3530 to 16596] | 13567.4 [7186 to 17164.4] | 10059.7 [5117 to 19944]
  Tumor necrosis factor receptor 1 (TNFR1) | 2007.2 [418.6 to 2593.2] | -77.2 [-161.7 to 604.6] | 6788 [793.1 to 34000.9] | 99.4 [-356.4 to 539.8]
  Tumor necrosis factor receptor 2 (TNFR2) | 8788 [3286 to 21126] | 75.4 [-693 to 4319] | 6788.2 [5440 to 14446] | -107.8 [-1726 to 1766]
  IL10 | 2.58 [1.66 to 7.77] | 2.58 [1.6 to 7.7] | 2.83 [1.31 to 4.93] | 2.6 [1.4 to 6.8]

ADVERSE EVENTS:
Arm/Group | Group 1: Thalidomide | Group 2: Placebo
Serious Adverse Events (participants affected / at risk) | 2/16 | 2/15
Other Adverse Events (participants affected / at risk) | 4/16 | 7/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Thalidomide (N=16) | Group 2: Placebo (N=15)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Drowsiness (Nervous system disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Thromboembolism (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Thalidomide (N=16) | Group 2: Placebo (N=15)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 5 (5)
Constipation (Gastrointestinal disorders) | 4 (4) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 5 (5)
Drowsiness (Nervous system disorders) | 4 (4) | 5 (5)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 4 (4) | 5 (5)
Numbness (Nervous system disorders) | 1 (1) | 6 (6)

LIMITATIONS AND CAVEATS:
Limited accrual and attrition led to small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No